CLINICAL TRIAL: NCT05387876
Title: Association of Vitamin D Supplementation and Normal Dietary Intake of Vitamin D With Changes in the Gut Microbiome and Markers of Colorectal Cancer Risk
Brief Title: Vitamin D Intervention and Associated Changes in the Gut Microbiome and Vitamin D Levels in Healthy Adults
Acronym: VDMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baylor University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BaylorU-VDMT
Record Dates: First submitted 2022-05-06; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled randomized intervention of vitamin supplementation
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators and outcomes assessors are masked to intervention group assignments using a researcher outside the study that maintains the study codes and IDs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo intervention (Placebo Comparator): A gummie candy the same consistency and nutrient value as the vitamin D gummie without any vitamin D will be taken as four gummies at the largest meal for 12 weeks once per day
  Interventions: Dietary Supplement: Placebo intervention
- Vitamin D intervention (Experimental): A vitamin D gummie the same consistency and nutrient value as the placebo gummie will be taken as four gummies at the largest meal for 12 weeks once per day providing 4000 IUs per day or 1000 IUs per gummie
  Interventions: Dietary Supplement: Vitamin D intervention

INTERVENTIONS:
Dietary Supplement: Vitamin D intervention — Nordic Naturals vitamin D gummies (1000 IUs/gummie), 4 gummies per day for 12 weeks
  Arms: Vitamin D intervention
Dietary Supplement: Placebo intervention — Organic gummie candies (no vitamin D), 4 gummies per day for 12 weeks
  Arms: Placebo intervention

SUMMARY:
Although dietary vitamin D supplementation has been used in the clinical setting for decades, the effect of supplementary vitamin D consumption on the structure of the microbiome has not been studied in humans in fine scale or with concomitant adjustment for dietary intake. Understanding the interaction of vitamin D with the microbiome in humans could lead to important advancements in the understanding of how vitamin D together with diet impacts the microbiome composition, and ultimately, risk of EOCRC. This study has the potential to lay the ground work for an adjunctive therapy to manipulate the microbiome to reduce risk of EOCRC. This proposed study is designed to evaluate the effect of vitamin D supplementation on the normal structure of the microbiome and data will not be used to diagnose, prevent, cure or treat disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years or older

Exclusion Criteria:

* Women who are currently pregnant or breastfeeding
* Use of antibiotics within the last 2 weeks
* Use of supplementary vitamin D within the last month
* Self-reported, pre-existing history of inflammatory bowel disease, heart disease or diabetes
* Students under 18
* Tanning/sun exposure > 60 min at a time in last 4 weeks
* No phenobarbital, carbamazepine, spironolactone chronic therapy; or steroid use within the last 2 weeks
* Severe allergy to ingredients found in supplements

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-12-03 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Microbiome alterations | 12 weeks
  Change in the microbiome structure and function

CONTACTS AND LOCATIONS:
Overall Officials: Kristen L Greathouse, PhD, Principal Investigator — Baylor University
Locations (1):
- Baylor University, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Study participant de-identified data will be shared with other researchers who submit a request for data acquisition. An MTA agreement will be constructed for protection of data sharing between the two researchers.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available at the time of publication in peer-reviewed journal for 10 years.
Access Criteria: Signed MTA agreement between study sponsor and requesting entity.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT05387876/Prot_SAP_000.pdf